CLINICAL TRIAL: NCT07094412
Title: Patient-engaged Development and Pilot Testing of Educational Content to Improve Understanding of Pharmacological vs Nocebo Effects of Statins
Brief Title: Patient-engaged Development and Testing of Educational Content on Side Effects of Statins
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-05028924
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dyslipidemia
Keywords: statin side effects; nocebo effect
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational intervention arm (Experimental): Participants view educational content
  Interventions: Other: Educational content on statin side effects

INTERVENTIONS:
Other: Educational content on statin side effects — Participants will view educational content that will include written material, graphics and video. The content will explain side effects and benefits of statin medications. The content will also explain placebo and nocebo effects and how they may impact people taking statins.

SUMMARY:
The purpose of this study is to learn about people's experiences and perspectives on side effects of statins and to use this information to develop and test educational content to help people understand statin side effects when they are newly prescribed a statin. Participants in the first phase of the study will fill out a survey and participate in a focus group or interview. Participants in the second phase of the study will view educational content, fill out a survey, and participate in two interviews.

ELIGIBILITY:
Inclusion Criteria:

* Has at least one cardiovascular risk factor, including diabetes (DM), hypertension (HTN), hyperlipidemia (HLD), or a 10-year risk of atherosclerotic cardiovascular disease (ASCVD) of equal to or greater than 7.5%
* Able to speak and read English

Exclusion Criteria:

* Established diagnosis of atherosclerotic cardiovascular disease (ASCVD), including coronary artery disease (CAD), peripheral arterial disease (PAD), or history of stroke
* Unable to access and engage with web-based education content for any reason (either independently or with the help of a support person)
* Is a healthcare professional at the college level or above, defined as a registered nurse, nurse practitioner, physician assistant, physician, dentist, or pharmacist
* Has a graduate-level degree of any kind
* Hospice or end-of-life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of educational intervention | Within 1 week of enrollment
  Number of enrolled participants who complete the educational intervention
Acceptability - satisfaction with educational intervention | Within 1 week of exposure to educational content
  Participants are asked to rate their satisfaction with the educational content on a scale of 1-5, ranging from 1-very dissatisfied to 5-very satisfied.
Acceptability - likelihood to recommend educational content | Within 1 week of exposure to the educational content
  Participants are asked how likely they are to recommend the educational content to friends or family, on a scale of 1 to 5, where 1 corresponds to "definitely will not recommend" and 5 corresponds to "definitely will recommend."

SECONDARY OUTCOMES:
Change in knowledge of statin side effects and benefits | At baseline, within 1 week of exposure to the educational content and again 4-6 weeks later
  Participants will be asked a series of questions (some multiple choice and some open-ended) about statin side effects and benefits. This instrument will be developed by the investigators during the first phase of the study which will utilize focus groups to explore patients experiences and beliefs with regard to statin side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Laura F Gingras, MD, MSc, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No